CLINICAL TRIAL: NCT06169267
Title: Phase III Intention to Treat Study of the Effect of Passive Music Intervention on Anxiety in Patients Undergoing Bone Marrow Aspiration and/or Biopsy
Brief Title: Passive Music Intervention for the Reduction of Anxiety in Patients Undergoing Bone Marrow Aspiration and/or Biopsy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22502; NCI-2023-09975 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22502 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm
MeSH Terms: interventions — Biopsy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (no music) (Active Comparator): Patients undergo standard of care bone marrow biopsy and/or aspiration.
  Interventions: Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Other: Questionnaire Administration
- Group II (listen to music) (Experimental): Patients listen to music while undergoing standard of care bone marrow biopsy and/or aspiration.
  Interventions: Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Music Therapy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration/biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration/biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Music Therapy — Listen to music
  Arms: Group II (listen to music)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of adding passive music when undergoing bone marrow biopsy/aspirate versus bone marrow biopsy/aspirate alone in reducing anxiety. Music therapy helps relieve pain or stress and promote well-being. Listening to music during a bone marrow biopsy/aspirate procedure may reduce anxiety during the procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether music listening alleviates psychological distress such as anxiety in patients undergoing bone marrow aspiration and/or biopsy that do not require general anesthesia.

SECONDARY OBJECTIVE:

I. To determine if patients with lower to no anxiety during bone marrow aspiration and/or biopsy will also experience less pain.

EXPLORATORY OBJECTIVE:

I. To design and implement an evidence-based music intervention protocol that could be used during bone marrow aspiration and/or biopsy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo standard of care bone marrow biopsy and/or aspiration.

GROUP II: Patients listen to music while undergoing standard of care bone marrow biopsy and/or aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Willingness to participate in the study
* Ability to read English, or willingness to have one of the staff members help with the questionnaire
* Age: ≥ 18 years
* Hematological conditions requiring a bone marrow biopsy and/or aspiration procedure, regardless of their disease state, and experience with such procedures

Exclusion Criteria:

* Hearing impairments, and non-verbal communication
* Scheduled to undergo a sedated bone marrow biopsy
* Scheduled to be premedicated with any anxiolytic or pain medication 30 minutes prior to the procedure
* Unwillingness to listen to music
* Altered mental health status that would prohibit informed consent and following protocol required instructions
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Changes in anxiety level | Up to 4 months
  Measured by State-Trait Anxiety Inventory (STAI) based on the response to 20 anxiety state-related questions, each scaled between 1 and 4, from low to high anxiety

SECONDARY OUTCOMES:
Pain level | Up to 4 months
  The visual analog scale ranging from 0 to 10 will be used to rate the pain level by subjects: 1-3 as mild, 4-6 as moderate and 7-10 as severe. The pain level will be compared between the music and non-music group by two-sample t tests. Univariate and multivariate analysis on pain level will be similar as that for anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States